CLINICAL TRIAL: NCT04875871
Title: Particle-based Partial Tumor Irradiation Targeting Hypoxic Segment and Sparing the Peritumoral Immune Microenvironment for Unresectable Bulky Tumors
Brief Title: Particle-based Partial Tumor Irradiation of Unresectable Bulky Tumors
Acronym: PARTICLE-PATHY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: targeted patient enrollment was not met.
Sponsor: EBG MedAustron GmbH (Industry)
Collaborators: Medical University of Vienna (Other); Landesklinkum Wiener Neustadt (Other); Klinik Ottakring (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PATHY-MA-072020
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: Particle Radiotherapy; Partial Tumor Irradiation
MeSH Terms: conditions — Neoplasms | interventions — Magnetic Resonance Imaging; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dose group (Experimental): 3 fractions of 12 Gy Relative Biological Effectiveness (RBE)
  Interventions: Radiation: Particle radiotherapy; Diagnostic Test: Magnetic resonance imaging; Diagnostic Test: Computertomography; Diagnostic Test: Copper-64-Diacetyl-bis (N4-methylthiosemicarbazone) Positron Emission Tomography-Computer Tomography (64Cu-ATSM-PET-CT); Diagnostic Test: 18-F-FluorDesoxyGlukose Positron Emission Tomography-Computer Tomography (18F-FDG-PET-CT); Diagnostic Test: Blood sampling
- Reduced-dose group (Experimental): 3 fractions of 8-10 Gy RBE
  Interventions: Radiation: Particle radiotherapy; Diagnostic Test: Magnetic resonance imaging; Diagnostic Test: Computertomography; Diagnostic Test: Copper-64-Diacetyl-bis (N4-methylthiosemicarbazone) Positron Emission Tomography-Computer Tomography (64Cu-ATSM-PET-CT); Diagnostic Test: 18-F-FluorDesoxyGlukose Positron Emission Tomography-Computer Tomography (18F-FDG-PET-CT); Diagnostic Test: Blood sampling

INTERVENTIONS:
Radiation: Particle radiotherapy — Partial radiotherapy targeting the hypoxic tumor segment
Diagnostic Test: Magnetic resonance imaging — For treatment planning as well as for follow-up radiological tumor assessment.
Diagnostic Test: Computertomography — For treatment planning as well as for follow-up radiological tumor assessment.
Diagnostic Test: Copper-64-Diacetyl-bis (N4-methylthiosemicarbazone) Positron Emission Tomography-Computer Tomography (64Cu-ATSM-PET-CT) — For the definition of the hypoxic tumor segment in treatment planning.
Diagnostic Test: 18-F-FluorDesoxyGlukose Positron Emission Tomography-Computer Tomography (18F-FDG-PET-CT) — For follow-up radiological tumor assessment.
Diagnostic Test: Blood sampling — Evaluation before treatment-start, during treatment and follow-up period.

SUMMARY:
This study uses a novel, recently developed unconventional radiotherapy technique which consists of three high-dose fractions directed to special segments of unresectable bulky tumors.

DETAILED DESCRIPTION:
This is a mono-centric, prospective, two-arms, feasibility study in which the investigator will enroll up to 22 patients with locally advanced or metastatic cancers with at least one bulky (≥6cm) lesion. This study uses a novel, recently developed unconventional radiotherapy technique, consisting of a short course (3 fractions) high dose partial irradiation targeting exclusively the hypoxic segment of unresectable bulky tumors while sparing the peritumoral immune microenvironment for induction of immune-mediated tumoricidal bystander and abscopal effects.

The present study will explore the potential biological and physical advantages of particle-based radiotherapy to deliver a highly conformal radiation dose to the hypoxic tumor segment defined by using hypoxia-specific Copper-64-Diacetyl-bis (N4-methylthiosemicarbazone) Positron Emission Tomography-Computer Tomography (64Cu-ATSM PET-CT) and dynamic contrast enhanced Magnetic Resonance Tomography imaging. Based on tumor location, volume and risk factors related to nearby organs at risk, patients will be divided in the "high-dose" or "reduced-dose" group which will be treated with different dose-schedules according to risk factors.

Additionally, radiotherapy will be administered at the precise timing, determined individually for each patient, based on the serially mapped homeostatic immune fluctuations by monitoring blood levels of the inflammatory markers. The objective is to synchronize the radiation treatment with the favorable, most reactive anti-tumor immune response phase, in order to break tumor´s immune-tolerance locally and systemically.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient prior to performing any treatment-related procedures.
2. Biopsy proven malignant unresectable solid bulky primary or recurrent tumor (diameter of at least 6 cm or greater, except for the Central Nervous System (CNS) tumors), or in a case of lack of recent biopsy progression on at least two consecutive radiological examinations, with biopsy proof in the past. Presence of locally advanced (cN+) and/or metastatic disease will be accepted in order to allow for assessment of the abscopal effects.
3. Ineligibility for standard treatments including surgery, conventional (whole tumor) radiotherapy and systemic therapy, or being in progression or stable (with no response to systemic treatment) under systemic therapy.
4. A minimum time interval from last dose of systemic therapy before radiotherapy of two weeks; Systemic therapy may be resumed 4 weeks following radiotherapy in order to permit assessment of the treatment efficacy.
5. Median life expectancy of >2 months.
6. Age > 18 years.
7. Adequate bone marrow function as follows below: Haemoglobin ≥ 8.0 g/d; Absolute neutrophil count (ANC) ≥ 1.5 x 10ꝰ/L (> 1500 per mm3); Platelet count ≥ 100 x 10ꝰ/L (>100,000 per mm3).
8. Female patients must either be of non-reproductive potential (i.e. post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) OR women of fertile age must have adequate conception prevention measures and must have a negative serum pregnancy test upon study entry.
9. Patient is willing and able to comply with the follow up including scheduled visits and examinations.

Exclusion Criteria:

1. Patients without bulky lesions.
2. Tumors suitable for the standard therapies including surgery, conventional (whole tumor) irradiation and systemic therapies.
3. Median life expectancy of less than 2 months.
4. Contraindication to i.v. Computer Tomography and Magnetic Resonance Tomography contrast medium administration, particularly estimated glomerular filtration rate (GFR) less than 45 mL/min/1.73 m2.
5. History of autoimmune disease.
6. Current or prior use of immunosuppressive medication within 14 days before enrollment with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
7. History of primary immunodeficiency.
8. History of allogeneic organ transplant.
9. Uncontrolled intercurrent comorbidity including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, active bleeding diatheses including any patient known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent.
10. Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control.
11. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results. (Note: criterion will be evaluated on the four eyes principle, evaluated by both Principle Investigator and Sub-Investigators.)
12. Patients with uncontrolled seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Bystander (local) tumor response rate | 11 months (after treatment)
  Bystander (local, at the level of the partially treated bulky tumor) response rate defined as at least a 30% regression of the unirradiated tumor tissue.

SECONDARY OUTCOMES:
Feasibility of PARTICLE-PATHY | 3,5 years (recruiting time + treatment time + 11 months follow-up)
  Feasibility of patient recruitment, treatment and follow-up rates.
Overall survival | 11 months (after treatment)
  Defined as the time from treatment until the time of death from any cause.
Time to local tumor progression | 11 months (after treatment)
  Defined as the time from treatment until the time of local disease progression.
Time to distant tumor progression | 11 months (after treatment)
  Defined as the time from treatment until the time of distant disease progression.
Abscopal (distant) tumor response rate | 11 months (after treatment)
  Defined as the proportion of metastatic patients that exhibited an abscopal effect versus the total number of metastatic patients allocated to the treatment.
Symptoms relief | 11 months (after treatment)
  Proportion of patients who will achieve a partial or complete relief at different time-points.
Radiation related toxicity | 11 months (after treatment)
  Toxicity assessment according to NCI CTCAE v5.0
Feasibility of timing of PARTICLE-PATHY and its relation to clinical outcomes | Until 11 months after treatment
  The feasibility of PARTICLE-PATHY and to it related TIMING will be defined by the proportion of patients allocated to this treatment who received it within dosimetric constraints after being able to define the immune-cycle periodicity and to synchronize radiotherapy with it versus the total number of patients allocated to the treatment.
Bystander/abscopal response rate in relation to dose-size of Peritumoral Immune Microenvironment (PIM) | 11 months (after treatment)
  See title
Bystander/abscopal response rate in relation to Interleukin-2 and Interferon Gamma values | 11 months (after treatment)
  Two key cytokines, Interleukin-2 (IL-2) and Interferon Gamma (INFg), will be serially assessed at baseline and after each radiotherapy treatment, in order to determine their potential role in modulating the immune response in relation to the bystander/abscopal effects.

CONTACTS AND LOCATIONS:
Overall Officials: Slavisa Tubin, M.D., Principal Investigator — EBG MedAustron
Locations (1):
- EBG MedAustron GmbH, Wiener Neustadt, Lower Austria, Austria